CLINICAL TRIAL: NCT02725450
Title: The Influence of Motor Imagery in Fine Motor Skills of Individuals With Disabilities
Brief Title: The Influence of Motor Imagery in Fine Motor Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Castelo Branco (Other)
Responsible Party: Principal Investigator, Pedro Alexandre Duarte Mendes, Phd, Instituto Politécnico de Castelo Branco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESE IPCB
Record Dates: First submitted 2016-03-23; First posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Mental Retardation and Developmental Disabilities With No Organic Condition
Keywords: Motor Imagery; Fine motor skills; Disabled
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motor Imagery + Psychomotor Battery of fine motor skills (Experimental): Application of Motor Imagery together with normal practice improves fine motor skills in disabled individuals.
  Interventions: Behavioral: Motor Imagery + Psychomotor Battery of fine motor skills; Behavioral: Psychomotor Battery of fine motor skills Practice

INTERVENTIONS:
Behavioral: Motor Imagery + Psychomotor Battery of fine motor skills — Subjects were randomly divided in two groups: a control group and an experimental one. The study procedures were applied on five different tasks of the Psychomotor Battery of fine motor skills (BPM). This instrument was applied in two stages, at the beginning of the study (pretest) and at the end of the 4 weeks (posttest). Both groups performed the tasks twice a week for a month. Motor imagery sessions were added on in the experimental group. Participants on the experimental group were asked to mentally imagine themselves recreating tasks they had performed earlier on the initial assessment.
Behavioral: Psychomotor Battery of fine motor skills Practice — Subjects were randomly divided in two groups: in the control group were applied on five different tasks of the Psychomotor Battery of fine motor skills (BPM). This instrument was applied in two stages, at the beginning of the study (pretest) and at the end of the 4 weeks (posttest). Both groups performed the tasks twice a week for a month.

SUMMARY:
The main purpose of this study is to ascertain whether the application of Motor Imagery together with normal practice improves fine motor skills in disabled individuals.

DETAILED DESCRIPTION:
Imagery is a cognitive process that can play an important role on the planning and execution of different movements or actions. The main purpose of this study is to ascertain whether the application of Motor Imagery together with normal practice improves fine motor skills in disabled individuals. In this study participated 42 subjects of both genders with disabilities, with a mean age of 37 (SD=12). Subjects were randomly divided in two groups: a control group and an experimental one. The study procedures were applied on five different tasks of the Psychomotor Battery of fine motor skills (BPM). This instrument was applied in two stages, at the beginning of the study (pretest) and at the end of the 4 weeks (posttest). Both groups performed the tasks twice a week for a month. Motor imagery sessions were added on in the experimental group. Participants on the experimental group were asked to mentally imagine themselves recreating tasks they had performed earlier on the initial assessment. For the analysis of the results, descriptive and inferential statistics were used. The T-test for independent samples, and the T-test for paired samples were applied.

ELIGIBILITY:
Inclusion Criteria:

* institutionalized individuals
* individuals with disabilities who were able to perform motor tasks

Exclusion Criteria:

* individuals with hearing disability
* individuals with visual disability
* individuals without motor autonomy

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Fine Motor Skill evaluated with Bateria Psicomotora (BPM) | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pedro AD Mendes, Phd, Principal Investigator — Instituto Politécnico de Castelo Branco

IPD SHARING:
Plan to Share IPD: Undecided